CLINICAL TRIAL: NCT00004814
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Copolymer 1 for Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Maryland (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/12023; UMB-55901
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Multiple Sclerosis; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Coat Protein Complex I

INTERVENTIONS:
Drug: copolymer 1

SUMMARY:
OBJECTIVES:

I. Compare tolerance to and therapeutic impact of copolymer 1, a mixture of synthetic polypeptides, with placebo in patients with relapsing-remitting multiple sclerosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution.

One group receives copolymer 1, a mixture of synthetic polypeptides composed of 4 amino acids, subcutaneously each day for 2 years.

The other group receives an injection of placebo daily for 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Clinically or laboratory-supported definite multiple sclerosis
* Neurologically stable for at least 30 days prior to entry Expanded Disability Status Scale score no greater than 5
* At least 2 documented relapses within 2 years prior to entry Onset of first relapse at least 1 year prior to randomization

--Prior/Concurrent Therapy--

* Biologic therapy: No prior copolymer 1
* Immunosuppressive therapy: No prior cytotoxic immunosuppressives, i.e.: Azathioprine Cyclophosphamide Cyclosporine At least 30 days since corticosteroids
* Radiotherapy: No prior lymphoid irradiation

--Patient Characteristics--

* Not HIV or HTLV-I seropositive No insulin-dependent diabetes mellitus No Lyme disease No requirement for aspirin or chronic nonsteroidal anti-inflammatory drugs No pregnant or nursing women Adequate contraception required of fertile women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250
Dates: Start 1991-10

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth P. Johnson, Study Chair — University of Maryland